CLINICAL TRIAL: NCT01767909
Title: Therapeutic Effects of Intranasally-Administered Insulin in Adults With Amnestic Mild Cognitive Impairment (aMCI) or Mild Alzheimer's Disease (AD)
Brief Title: The Study of Nasal Insulin in the Fight Against Forgetfulness (SNIFF)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Alzheimer's Therapeutic Research Institute (Other); Wake Forest University Health Sciences (Other)
Responsible Party: Principal Investigator, Paul S. Aisen, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADC-046-INI; RF1AG041845 (NIH)
Record Dates: First submitted 2013-01-10; First posted 2013-01-15 (Estimated); Results first posted 2020-05-18 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Amnestic Mild Cognitive Impairment; Alzheimer's Disease
Keywords: Intranasal insulin; Alzheimer's disease; Amnestic mild cognitive impairment; Dementia; Brain diseases; Memory problems; Mental disorders; Cognitive disorders
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Memory Disorders; Mental Disorders; Cognitive Dysfunction | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin (Humulin® R U-100) (Experimental): 120 subjects will take two daily doses of INI (20 IU bid for a total daily dose of 40 IU) approximately 30 minutes after breakfast and dinner for 12 months. A 6-month open label period will follow in which all participants will receive INI.
  Interventions: Drug: Insulin (Humulin® R U-100)
- Placebo (Placebo Comparator): 120 subjects will take two daily doses of placebo approximately 30 minutes after breakfast and dinner for 12 months. A 6-month open label period will follow in which all participants will receive INI.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Insulin (Humulin® R U-100) — 20 IU bid taken twice daily (approximately 30 minutes after breakfast and dinner) for a total of 40 IU daily, which will be administered intranasally. The device used to administer insulin releases a metered dose into a chamber covering the participant's nose. The insulin is then inhaled by breathing evenly over a specified period.
  Arms: Insulin (Humulin® R U-100)
Drug: Placebo — Placebo taken twice daily (approximately 30 minutes after breakfast and dinner), which will be administered intranasally. The device used to administer placebo releases a metered dose into a chamber covering the participant's nose. The placebo is then inhaled by breathing evenly over a specified period.
  Arms: Placebo

SUMMARY:
An urgent need exists to find effective treatments for Alzheimer's disease (AD) that can arrest or reverse the disease at its earliest stages. The emotional and financial burden of AD to patients, family members, and society is enormous, and is predicted to grow exponentially as the median population age increases. Current FDA-approved therapies are modestly effective at best. This study will examine a novel therapeutic approach using intranasal insulin (INI) that has shown promise in short-term clinical trials. If successful, information gained from the study has the potential to move INI forward rapidly as a therapy for AD. The study will also provide evidence for the mechanisms through which INI may produce benefits by examining key cerebral spinal fluid (CSF) biomarkers and hippocampal/entorhinal atrophy. These results will have considerable clinical and scientific significance, and provide therapeutically-relevant knowledge about insulin's effects on AD pathophysiology. Growing evidence has shown that insulin carries out multiple functions in the brain, and that insulin dysregulation may contribute to AD pathogenesis.

This study will examine the effects of intranasally-administered insulin on cognition, entorhinal cortex and hippocampal atrophy, and cerebrospinal fluid (CSF) biomarkers in amnestic mild cognitive impairment (aMCI) or mild AD. It is hypothesized that after 12 months of treatment with INI compared to placebo, subjects will improve performance on a global measure of cognition, on a memory composite and on daily function. In addition to the examination of CSF biomarkers and hippocampal and entorhinal atrophy, the study aims to examine whether baseline AD biomarker profile, gender, or Apolipoprotein epsilon 4 (APOE-ε4) allele carriage predict treatment response.

In this study, 240 people with aMCI or AD will be given either INI or placebo for 12 months, following an open-label period of 6 months where all participants will be given active drug. The study uses insulin as a therapeutic agent and intranasal administration focusing on nose to brain transport as a mode of delivery.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English or Spanish
* Diagnosis of aMCI by Petersen criteria or probable AD by National Institute of Neurological and Communicative Diseases and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria
* Mini Mental State Examination (MMSE) score at screening is greater than or equal to 20
* Clinical Dementia Rating is 0.5-1 at screening
* Logical Memory is less than or equal to 8 for 16 or more years of education, less than or equal to 4 for 8-15 years of education, less than or equal to 2 for 0-7 years of education. Scores measured at screening on Delayed Paragraph Recall (Paragraph A only) from the Wechsler Memory Scale-Revised
* Able to complete baseline assessments
* Modified Hachinski score of less than or equal to 4
* A study partner able to accompany the participant to most visits and answer questions about the participant
* The study partner must have direct contact with the participant more than 2 days per week (minimum of 10 hours per week) and provide supervision of drug administration as needed
* Stable medical condition for 3 months prior to screening visit
* Stable medications for 4 weeks prior to the screening and baseline visits
* Stable use of permitted medications
* At least six years of education or work history
* Clinical laboratory values must be within normal limits or, if abnormal, must be judged to be clinically insignificant by the investigator
* Visual and auditory acuity adequate for neuropsychological testing

Exclusion Criteria:

* A diagnosis of dementia other than probable AD
* Probable AD with Down syndrome
* History of clinically significant stroke
* Current evidence or history in past two years of epilepsy, focal brain lesion, head injury with loss of consciousness or Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM IV) criteria for any major psychiatric disorder including psychosis, major depression, bipolar disorder, alcohol or substance abuse
* Sensory impairment that would preclude the participant from participating in or cooperating with the protocol
* Diabetes (type 1 or type II) requiring pharmacologic treatment (including both insulin dependent and non-insulin dependent diabetes mellitus)
* Current or past use of insulin or any other anti-diabetic medication
* Evidence of any significant clinical disorder or laboratory finding that renders the participant unsuitable for receiving investigational drug including clinically significant or unstable hematologic, hepatic, cardiovascular, pulmonary, endocrine, metabolic, renal or other systemic disease or laboratory abnormality.
* Active neoplastic disease, history of cancer five years prior to screening (history of skin melanoma or stable prostate cancer are not excluded)
* History of seizure within the past five years
* Pregnancy or possible pregnancy
* Contraindications to Lumbar Puncture (LP) procedure: prior lumbosacral spine surgery, severe degenerative joint disease or deformity of the spine, platelets is less than 100,000 or history of bleeding disorder
* Use of anticoagulants warfarin (Coumadin) and dabigatran (Pradaxa) due to LP requirement
* Contraindications for MRI (claustrophobia, craniofacial metal implants of any kind, pacemakers)
* Residence in a skilled nursing facility at screening
* Use of an investigational agent within two months or screening visit
* Regular use of narcotics, anticonvulsants, medications with significant anticholinergic activity, antiparkinsonian medications or any other exclusionary medications

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2014-01-08 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2018-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Craft, PhD, Study Director — Wake Forest University Health Sciences; Paul Aisen, MD, Study Director — USC Alzheimer's Therapeutic Research Institute (ATRI)
Locations (25):
- United States (25):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Barrow Neurology Clinics, Phoenix, Arizona
  - University of California, Irvine, Irvine, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Howard University, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Mount Sinai School of Medicine, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Case Western Reserve University, Beachwood, Ohio
  - Tulsa Clinical Research, Tulsa, Oklahoma
  - Rhode Island Hospital, Providence, Rhode Island
  - Roper St. Francis Hospital, Charleston, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - U of WA / VA Puget Sound Alzheimer's Disease Research Center, Seattle, Washington

REFERENCES:
- [Background] Craft S, Baker LD, Montine TJ, Minoshima S, Watson GS, Claxton A, Arbuckle M, Callaghan M, Tsai E, Plymate SR, Green PS, Leverenz J, Cross D, Gerton B. Intranasal insulin therapy for Alzheimer disease and amnestic mild cognitive impairment: a pilot clinical trial. Arch Neurol. 2012 Jan;69(1):29-38. doi: 10.1001/archneurol.2011.233. Epub 2011 Sep 12. PMID 21911655
- [Background] Craft S, Peskind E, Schwartz MW, Schellenberg GD, Raskind M, Porte D Jr. Cerebrospinal fluid and plasma insulin levels in Alzheimer's disease: relationship to severity of dementia and apolipoprotein E genotype. Neurology. 1998 Jan;50(1):164-8. doi: 10.1212/wnl.50.1.164. PMID 9443474
- [Background] Reger MA, Watson GS, Green PS, Wilkinson CW, Baker LD, Cholerton B, Fishel MA, Plymate SR, Breitner JC, DeGroodt W, Mehta P, Craft S. Intranasal insulin improves cognition and modulates beta-amyloid in early AD. Neurology. 2008 Feb 5;70(6):440-8. doi: 10.1212/01.WNL.0000265401.62434.36. Epub 2007 Oct 17. PMID 17942819
- [Background] Baker LD, Cross DJ, Minoshima S, Belongia D, Watson GS, Craft S. Insulin resistance and Alzheimer-like reductions in regional cerebral glucose metabolism for cognitively normal adults with prediabetes or early type 2 diabetes. Arch Neurol. 2011 Jan;68(1):51-7. doi: 10.1001/archneurol.2010.225. Epub 2010 Sep 13. PMID 20837822
- [Derived] Donohue MC, Langford O, Insel PS, van Dyck CH, Petersen RC, Craft S, Sethuraman G, Raman R, Aisen PS; Alzheimer's Disease Neuroimaging Initiative. Natural cubic splines for the analysis of Alzheimer's clinical trials. Pharm Stat. 2023 May-Jun;22(3):508-519. doi: 10.1002/pst.2285. Epub 2023 Jan 10. PMID 36627206
- [Derived] Kellar D, Lockhart SN, Aisen P, Raman R, Rissman RA, Brewer J, Craft S. Intranasal Insulin Reduces White Matter Hyperintensity Progression in Association with Improvements in Cognition and CSF Biomarker Profiles in Mild Cognitive Impairment and Alzheimer's Disease. J Prev Alzheimers Dis. 2021;8(3):240-248. doi: 10.14283/jpad.2021.14. PMID 34101779
- [Derived] Craft S, Raman R, Chow TW, Rafii MS, Sun CK, Rissman RA, Donohue MC, Brewer JB, Jenkins C, Harless K, Gessert D, Aisen PS. Safety, Efficacy, and Feasibility of Intranasal Insulin for the Treatment of Mild Cognitive Impairment and Alzheimer Disease Dementia: A Randomized Clinical Trial. JAMA Neurol. 2020 Sep 1;77(9):1099-1109. doi: 10.1001/jamaneurol.2020.1840. PMID 32568367
- See also: Alzheimer's Therapeutic Research Institute (ATRI) — http://keck.usc.edu/atri/research/studies/

RESULTS

PARTICIPANT FLOW:
Groups:
- Insulin (Humulin® R U-100): 20 IU BID intranasal insulin (Humulin® R U-100) twice daily for a total of 40 IU daily for 12 months, followed by a 6-month open label period.
- Placebo: 50% of participants received placebo treatment twice daily for 12 months followed by a 6-month open label period where all participants received 20 IU BID intranasal insulin (Humulin® R U-100) twice daily (total of 40 IU daily).
Period: Overall Study
Arm/Group | Insulin (Humulin® R U-100) | Placebo
Started | 121 | 119
Completed | 108 | 107
Not Completed | 13 | 12
Not completed — Withdrawal by Subject | 4 | 7
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Study Partner | 3 | 1
Not completed — Non-Compliance | 2 | 0
Not completed — Perceived Lack of Efficacy | 1 | 0
Not completed — Investigator Recommendation | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — LP uncessessful | 0 | 1

BASELINE CHARACTERISTICS:
Population: This represents the final baseline characteristics report for the blinded phase of the INI study. Population: Intent-To-Treat [ITT] population: All randomized participants in Impel Device.
Groups:
- Insulin (Humulin® R U-100): 50% of participants received 20 IU BID intranasal insulin (Humulin® R U-100) twice daily for a total of 40 IU daily for 12 months, followed by a 6-month open label period.
- Total: Total of all reporting groups
Arm/Group | Insulin (Humulin® R U-100) | Placebo | Total
Number analyzed (Participants) | 121 | 119 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.46 (7.38) | 71.06 (6.79) | 70.76 (7.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 58 | 117
  Male | 62 | 61 | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 116 | 113 | 229
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 117 | 108 | 225
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Education [Mean (Standard Deviation); unit: years] | 16.07 (2.64) | 16.31 (2.92) | 16.19 (2.78)
ApoE-e4 carrier status (Positive vs Negative) [Count of Participants; unit: Participants]
  Negative | 42 | 42 | 84
  Positive | 79 | 77 | 156
Alzheimer's Disease Assessment Scale-Cognitive 12 (ADAS-Cog12) [Mean (Standard Deviation); unit: units on a scale] — The ADAS-Cog is a psychometric instrument that evaluates memory, attention, reasoning, language, orientation, and praxis. The ADAS-Cog12 version was used in this study which includes Delayed Word Recall - a measure of episodic memory. Scores from the original portion of the test range from 0 (best) to 70 (worse) and then number of items not recalled ranging from 0-10 is added for a maximum score of 80. A higher score indicates more impairment. Population: Number of participants analyzed is lower than the total number of baselined participants due to the primary analysis being a modified intent-to-treat (mITT) analysis using the mixed model repeated measures (MMRM) where only randomized participants with at least one post-baseline assessment are included.
  units on a scale
    number analyzed (Participants) | 121 | 118 | 239
    (all) | 25.91 (8.28) | 24.73 (7.56) | 25.33 (7.94)
Clinical Dementia Rating Scale - Sum of Boxes (CDR-SB) [Mean (Standard Deviation); unit: units on a scale] — The CDR-SB is administered as a structured interview with the participant and study partner, where impairment is scored in each of 6 categories: memory, orientation, judgment and problem solving, community affairs, home and hobbies and personal care. Impairment is scored on a scale in which none = 0, questionable = 0.5, mild = 1, moderate = 2 and severe = 3. The 6 individual category ratings, or "box scores", are added together to give the CDR-Sum of Boxes which ranges from 0-18 with higher scores indicated more impairment.
  units on a scale | 3.59 (1.51) | 3.35 (1.51) | 3.47 (1.51)
Memory Composite (Story Recall and the Free and Cued Selective Reminding Test) [Mean (Standard Deviation); unit: units on a scale] — This study used a Memory Composite composed of Story Recall (Immediate and Delayed), and Free and Cued Selective Reminding Test. Each of the three component scores were normalized by subtracting the baseline sample mean, and dividing by the baseline sample standard deviation, to form three separately standardized z-scores with mean 0 and standard deviation 1. The three Z-scores were summed to form the memory composite. No other standardization was performed on the sum. In this study, the composite scores ranged from about -4.74 to 9.15 at baseline. A higher score indicates better performance. Population: Number of participants analyzed is lower than the total number of baselined participants due to the primary analysis being a modified intent-to-treat (mITT) analysis using the mixed model repeated measures (MMRM) where only randomized participants with at least one post-baseline assessment are included.
  units on a scale
    number analyzed (Participants) | 117 | 113 | 230
    (all) | -0.16 (2.47) | 0.25 (2.59) | 0.04 (2.53)

OUTCOME MEASURES:

1. Primary Outcome: Change in Global Measure of Cognition as Measured by the Alzheimer's Disease Assessment Scale-Cognitive 12 (ADAS-Cog12)
Description: The ADAS-Cog is a psychometric instrument that evaluates memory, attention, reasoning, language, orientation, and praxis. The ADAS-Cog12 version was used in this study which includes Delayed Word Recall - a measure of episodic memory. Scores from the original portion of the test range from 0 (best) to 70 (worse) and then number of items not recalled ranging from 0-10 is added for a maximum score of 80. A positive change indicates cognitive worsening.
Time Frame: 12 months (blinded phase) followed by 6 months (open label phase)
Population: Modified intent-To-Treat [mITT] population: All randomized participants in Impel Device with ADAS-Cog12 observed at baseline and at least one follow-up.
Measure: Least Squares Mean (Standard Error); unit: Modeled change score on a scale
Arm/Group | Insulin (Humulin® R U-100) | Placebo
Number analyzed (Participants) | 121 | 119
Modeled change score on a scale
  Blinded Phase (M12 change from Baseline) | 3.893 (0.643) | 3.867 (0.650)
  Open Label Phase (M18 change from Baseline) | 7.091 (0.937) | 6.164 (0.942)

2. Secondary Outcome: Change in Memory Composite as Measured by Story Recall (Immediate Paragraph Recall and Delayed Paragraph Recall) and Free and Cued Selective Reminding Test (FCSRT)
Description: Memory Composite is composed from Story Recall (both Immediate Paragraph Recall and Delayed Paragraph Recall) and the Free and Cued Selective Reminding Test (FCSRT). Each of the three component scores were normalized by subtracting the baseline sample mean, and dividing by the baseline sample standard deviation, to form three separately standardized z-scores with mean 0 and standard deviation 1. The three Z-scores were summed to form the memory composite. No other standardization was performed on the sum. If any of Immediate Paragraph Recall, Delayed Paragraph Recall and FCSRT is missing, the memory composite is missing. Higher scores indicate better performance. In this study the scores ranged from about -4.74 to 9.15 at baseline, and about -5.10 to 9.43 across all visits over 12 months.
Time Frame: 12 months (blinded phase) followed by 6 months (open label phase)
Measure: Least Squares Mean (Standard Error); unit: modeled change score on a scale
Arm/Group | Insulin (Humulin® R U-100) | Placebo
Number analyzed (Participants) | 121 | 119
modeled change score on a scale
  Blinded Phase (M12 change from Baseline) | -0.496 (0.163) | -0.433 (0.162)
  Open Label Phase (M18 change from Baseline) | -0.594 (0.183) | -0.802 (0.184)

3. Secondary Outcome: Change in Daily Functioning as Measured by the ADCS-MCI Activities of Daily Living (ADCS-ADL-MCI)
Description: The Alzheimer's Disease Cooperative Study - Activities of Daily Living Scale (ADCS-ADL) is an activities of daily living questionnaire aimed at detecting functional decline in people with Mild Cognitive Impairment (MCI). In a structured interview format, informants are queried as to whether participants attempted each item in the inventory during the prior 4 weeks and their level of performance. The questions focus predominantly on instrumental activities of daily living scales (e.g. shopping, preparing meals, using household appliances, keeping appointments, reading). The total score can range from 0-54. A higher score indicates greater functional ability.
Time Frame: 12 months (blinded phase) and 6 months (open label phase)
Population: Modified intent-To-Treat [mITT] population: All randomized participants in Impel Device with ADCS-ADL-MCI observed at baseline and at least one follow-up.
Measure: Least Squares Mean (Standard Error); unit: modeled change score on a scale
Arm/Group | Insulin (Humulin® R U-100) | Placebo
Number analyzed (Participants) | 121 | 119
modeled change score on a scale
  Blinded Phase (M12 change from Baseline) | -3.63 (0.769) | -4.26 (0.779)
  Open Label Phase (M18 change from baseline) | -7.35 (0.925) | -6.56 (0.934)

4. Secondary Outcome: Change in Cognitive Deficit as Measured by Clinical Dementia Rating - Sum of Boxes (CDR-SB)
Description: The Clinical Dementia Rating - Sum of Boxes (CDR-SB) is administered as a structured interview with the participant and study partner, where impairment is scored in each of categories: memory, orientation, judgment and problem solving, community affairs, home and hobbies and personal care. Impairment is scored on a scale in which none = 0, questionable = 0.5, mild = 1, moderate = 2 and severe = 3. The 6 individual category ratings, or "box scores", are added together to give the CDR-Sum of Boxes which ranges from 0-18 with higher scores indicated more impairment.
Time Frame: 12 months (blinded phase) followed by 6 months (open label phase)
Population: Modified intent-To-Treat [mITT] population: All randomized participants in Impel Device with CDR-SB observed at screening and at least one follow-up.
Measure: Least Squares Mean (Standard Error); unit: Modeled change in test score
Arm/Group | Insulin (Humulin® R U-100) | Placebo
Number analyzed (Participants) | 121 | 119
Modeled change in test score
  Blinded Phase (M12 change from Baseline) | 1.682 (0.195) | 1.402 (0.196)
  Open Label Phase (M18 change from Baseline) | 2.361 (0.247) | 2.122 (0.249)

5. Secondary Outcome: Change in Hippocampal and Entorhinal Atrophy as Measured by Magnetic Resonance Imaging (MRI)
Description: MRI will be used to assess the effect of treatment on rate of hippocampal and entorhinal atrophy, and conduct exploratory analyses of other brain regions. Volume change was normalized to the participant's own intracranial volume to account for each participant's brain size.
Time Frame: Screen and Month 12
Population: Intent-To-Treat [ITT] population: All randomized participants in Impel Device. Follow-up visits include month 12 and early termination 1 (et1) visits. Percent change data is available for 3 subjects with et1 visit and 187 subjects with month 12 as follow-up.
Measure: Mean (Standard Deviation); unit: % change in volume
Arm/Group | Insulin (Humulin® R U-100) | Placebo
Number analyzed (Participants) | 116 | 116
% change in volume
  Normalized hippocampal volume change | -0.01 (0.02) | -0.02 (0.02)
  Normalized entorhinal volume change | -0.01 (0.03) | -0.01 (0.03)
  Normalized whole brain volume change | -1.35 (1.09) | -1.41 (1.18)

6. Secondary Outcome: Change in CSF Biomarkers of AD
Description: Quantify Abeta and Tau biomarkers in CSF
Time Frame: Baseline and Month 12
Population: CSF collection was optional; only a subset of participants underwent the LP procedure
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Insulin (Humulin® R U-100) | Placebo
Number analyzed (Participants) | 72 | 75
pg/ml
  Abeta 40 | -264.851 (1168.995) | -127.539 (1600.604)
  Abeta 42 | -15.552 (61.884) | -4.456 (82.156)
  Total Tau | -4.717 (263.810) | 1.937 (291.160)
  p-Tau | -2.764 (18.729) | -0.567 (25.293)

ADVERSE EVENTS:
Time Frame: Adverse Event Table represents data collected over a period of 12 months (blinded phase).
Description: "Other (Not Including Serious) Adverse Events" reported include both Serious and Non Serious Adverse Events.
Arm/Group | Insulin (Humulin® R U-100) | Placebo
All-Cause Mortality (participants affected / at risk) | 1/121 | 0/119
Serious Adverse Events (participants affected / at risk) | 18/121 | 10/119
Other Adverse Events (participants affected / at risk) | 98/121 | 91/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin (Humulin® R U-100) (N=121) | Placebo (N=119)
BLOOD AND LYMPHATIC SYSTEM DISORDERS (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
CARDIAC DISORDERS (Cardiac disorders) | 2 (2) | 3 (4)
GASTROINTESTINAL DISORDERS (Gastrointestinal disorders) | 3 (3) | 1 (1)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS (General disorders) | 1 (3) | 2 (2)
HEPATOBILIARY DISORDERS (Hepatobiliary disorders) | 1 (1) | 0 (0)
INFECTIONS AND INFESTATIONS (Infections and infestations) | 1 (1) | 2 (2)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
NERVOUS SYSTEM DISORDERS (Nervous system disorders) | 1 (1) | 2 (2)
PSYCHIATRIC DISORDERS (Psychiatric disorders) | 1 (1) | 0 (0)
RENAL AND URINARY DISORDERS (Renal and urinary disorders) | 2 (3) | 0 (0)
VASCULAR DISORDERS (Vascular disorders) | 4 (7) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin (Humulin® R U-100) (N=121) | Placebo (N=119)
BLOOD AND LYMPHATIC SYSTEM DISORDERS (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
CARDIAC DISORDERS (Cardiac disorders) | 8 (9) | 6 (8)
DEMENTIA AND AMNESTIC CONDITIONS (Nervous system disorders) | 0 (0) | 1 (1)
ENDOCRINE DISORDERS (Endocrine disorders) | 1 (1) | 0 (0)
EYE DISORDERS (Eye disorders) | 5 (5) | 2 (2)
GASTROINTESTINAL DISORDERS (Gastrointestinal disorders) | 21 (26) | 13 (17)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS (General disorders) | 11 (11) | 7 (8)
HEPATOBILIARY DISORDERS (Hepatobiliary disorders) | 1 (1) | 0 (0)
IMMUNE SYSTEM DISORDERS (Immune system disorders) | 2 (2) | 1 (1)
INFECTIONS AND INFESTATIONS (Infections and infestations) | 32 (36) | 27 (32)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS (Injury, poisoning and procedural complications) | 20 (31) | 30 (36)
INVESTIGATIONS (Investigations) | 6 (9) | 4 (4)
METABOLISM AND NUTRITION DISORDERS (Metabolism and nutrition disorders) | 4 (6) | 4 (5)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS (Musculoskeletal and connective tissue disorders) | 17 (20) | 16 (19)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (10) | 6 (6)
NERVOUS SYSTEM DISORDERS (Nervous system disorders) | 19 (23) | 21 (25)
PSYCHIATRIC DISORDERS (Psychiatric disorders) | 18 (20) | 20 (23)
RENAL AND URINARY DISORDERS (Renal and urinary disorders) | 7 (8) | 3 (3)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS (Respiratory, thoracic and mediastinal disorders) | 20 (23) | 24 (28)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS (Skin and subcutaneous tissue disorders) | 10 (11) | 6 (6)
SURGICAL AND MEDICAL PROCEDURES (Surgical and medical procedures) | 2 (3) | 1 (1)
VASCULAR DISORDERS (Vascular disorders) | 15 (20) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs agree to provide a copy of the manuscript to Dr. Suzanne Craft, Project Director, Wake Forest School of Medicine, and the National Institutes of Health (NIH) must be cited as a funding agency.

DOCUMENTS (2):
  • Study Protocol (2016-12-05): https://cdn.clinicaltrials.gov/large-docs/09/NCT01767909/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT01767909/SAP_001.pdf